CLINICAL TRIAL: NCT04624373
Title: Molecular Analysis of the Surnantant of Echoguidated Bronchoscopic Cytopunctions in Lung Cancer
Brief Title: Genotyping of Ebus-tbna Supernant Cell-free Dna in Nsclc
Acronym: CELTICS
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/19/0090
Record Dates: First submitted 2020-11-09; First posted 2020-11-10 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Lung Cancer
Keywords: NSCLC; genotyping; liquid biopsy; cytology supernatant
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Identified mutation: The sensitivity of supernatant to identify the mutations detected on cell block (Gold standard).
  Interventions: Other: Molecular analysis of surnatant
- Non identified mutation: The sensitivity of supernatant to identify the mutations detected on cell block (Gold standard).
  Interventions: Other: Molecular analysis of surnatant

INTERVENTIONS:
Other: Molecular analysis of surnatant — The interventional pulmonologist selects the most suspect node. The corresponding TBNA is placed in Cytolyt and tagged using a sticker to indicate the specimen from which supernatant must be saved after the initial spin.
  The supernatant is transferred to the "Laboratoire de Biologie Médicale Oncologique" where it undergoes a further hard spin. The remaining supernatant is stored at -80°C before to send it to Foundation One for DNA extraction from 3 ml of supernatant and genotyping.
  Two 7,5 mL blood tubes are transferred to the laboratory to extract plasma. Plasma was stored at -80°C and then sent to Foundation One for DNA extraction from 2 mL of plasma and genotyping.
  10 slides from the cell block are shipped to Foundation One. These specimens are tested by FoundationOne®CDX (tissue), and FoundationOne®Liquid (supernatant and plasma) for genomic and TMB analyses (hybrid-capture based next generation sequencing).

SUMMARY:
The wide uptake of "liquid biopsy" diagnostics in the care of advanced cancer patients highlights the desire for improved access to tumor allowing accurate tumor genotyping (1). Genotyping of plasma cfDNA is now routine for detection of EGFR driver mutations at diagnosis of NSCLC, or for detection of the EGFR T790M mutation after TKI resistance, and is an emerging approach for the detection of other drivers (HER2 or BRAF mutations, ALK or ROS1 fusions…) (2) or the estimation of tumor mutation burden (TMB) (3). However, the most sensitive plasma genotyping platforms still have a sensitivity of only 70%-80%, such that a negative result requires tissue biopsy confirmation.

DETAILED DESCRIPTION:
The wide uptake of "liquid biopsy" diagnostics in the care of advanced cancer patients highlights the desire for improved access to tumor allowing accurate tumor genotyping (1). Genotyping of plasma cfDNA is now routine for detection of EGFR driver mutations at diagnosis of NSCLC, or for detection of the EGFR T790M mutation after TKI resistance, and is an emerging approach for the detection of other drivers (HER2 or BRAF mutations, ALK or ROS1 fusions…) (2) or the estimation of tumor mutation burden (TMB) (3). However, the most sensitive plasma genotyping platforms still have a sensitivity of only 70%-80%, such that a negative result requires tissue biopsy confirmation. This poses a clinical challenge because negative plasma genotyping is correlated with more limited metastatic spread and lower tumor burden, such that biopsy of these patients may be even more challenging. Because invasive biopsy remains an integral part of the diagnostic strategy, methods are needed for maximizing the yield from these biopsy procedures.

There is a current paradox between the need for large amounts of tissue for multiplex analysis of an increasing number of targetable drivers and markers of response to immune therapy (PD-L1, TMB) and the development of minimally invasive biopsy procedures that results in limited specimens. Up to 25% of patients are thus treated without knowledge of the molecular profile of their tumor (4). In particular, 20% of endobronchial ultrasonography transbronchial needle aspiration (EBUS-TBNA) are rejected from genotyping due to lack of tissue (5) after time and tissue consuming diagnostics steps that are sometimes not required (resistance setting). Circulating tumor DNA is an emerging approach for cancer genotyping but sensitivity is limited to 70-80% (6) by inconsistent tumor shed and low DNA concentrations, so that tissue biopsy is still routine. Also, feasibility of TMB assessment on tissue is only 60% (likely much less on EBUS-TBNA specimens) (7) and approximately 80% in plasma (blood TMB, bTMB) (3).

The presence of cfDNA in several biological fluids and the feasibility of detecting mutations of interest (usually targeting only EGFR) in these fluids (urine, pleural fluid, CSF) have been clearly demonstrated (8-12), while blood is the most widely studied liquid biopsy substrate in advanced NSCLC.

Furthermore, we showed in a proof of concept study, investigating various FNA specimens in a limited numbers of patients that cytology samples' supernatant (usually discarded) is a rich source of DNA. Our results suggest that supernatant free DNA (sfDNA) can be used for baseline and resistance genotyping (13).

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years-old
* Patients planned for an EBUS-TBNA for

  1. Suspicion of stage IV lung cancer (PET+ mediastinal node(s)) (Cohort 1)
  2. Stage IV NSCLC with an EGFR, BRAF, HER2, MET mutation or ALK, RET or ROS1 rearranged NSCLC and acquired resistance to targeted therapy (Cohort 2)
* Performance status 0-3
* Informed consent

Exclusion Criteria:

* Refusal to participate
* Patient under legal tutelage

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited in our Department in Toulouse University Hospital, during appointment needed for information and planning of the EBUS-TBNA procedure.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
main aim of the study | 18 months
  to investigate the sensitivity of sfDNA genotyping in various clinical settings and to compare it to cell block

SECONDARY OUTCOMES:
TMB estimation | 18 months
  To assess the feasibility of TMB estimation on this specimen
sensitivity of plasma | 18 months
  To compare the sensitivity of plasma genotyping to cell block
concordance between plasma and supernatant | 18 months
  To investigate the concordance between plasma and supernatant for mutation detection and TMB estimation
mutation rate | 18 months
  To calculate the rate of patients with at least one additional mutation detected on supernatant compared to cell block
Sensitivity of supernatant and plasma | 18 months
  To compare the sensitivity of supernatant and plasma to cell block for the detection of specific alterations (EGFR, HER2, BRAF, PIK3CA, KRAS, MET mutations, ALK, ROS1, NTRK, RET fusions)
Turnaround time of supernatant | 18 months
  To compare the turnaround time of supernatant, plasma and cell block for genotyping

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Guibert, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Nicolas Guibert, Toulouse, France